CLINICAL TRIAL: NCT06400875
Title: A Prospective, Multi Center Observational Study to Investigate the Safety and Effectiveness of Sterilized, Porcine Placental Tissue in the Treatment of Chronic Venous Leg Ulcers
Brief Title: Observational Study to Investigate the Use of Sterilized Porcine Placental Tissue in the Treatment of Chronic VLU
Status: Active, not recruiting | Type: Observational
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TLS-IM-002
Record Dates: First submitted 2024-04-27; First posted 2024-05-06 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Ulcer Venous; Wound Heal
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: InnovaMatrix® AC Sterilized, Porcine Placental Extracellular Matrix (ECM) — weekly application of sterilized, porcine placental ECM followed by standard of care wound therapy and compression therapy

SUMMARY:
The study is a multi-center, prospective, clinical trial designed to evaluate the use of InnovaMatrix AC sterilized porcine placental ECM to treat chronic VLUs . The trial will include 30 completed subjects at multiple, experienced clinical centers in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients over 18 years of age who have given written informed consent in accordance with the ICH Good Clinical Practice (GCP) guideline. Female subjects must be either of non-childbearing potential or if of childbearing potential must satisfy the defined contraceptive criteria Exclusion criteria.
2. Patients who are willing and able to attend all follow-up visits.
3. Index ulcer characteristics:

   1. Ulcer present for ≥ 30 days prior to (Day 0).
   2. Index ulcer is above the malleolus.
   3. Ulcer greater than or equal to 2cm2 and less than or equal to 20cm2 at the time of enrollment.
4. Subject has adequate circulation to the affected extremity, as demonstrated by at least one of the following within the past 30 days:

   * Dorsum transcutaneous oxygen test (TcPO2) with results ≥ 30 mmHg, Or
   * ABIs with results of ≥ 0.7 and ≤ 1.2, Or
   * Doppler arterial waveforms, which are triphasic or biphasic at the ankle of the affected foot. For ABPI >1.2 TBI (Toe Brachial Index) > 0.5.
   * Patient able to ambulate at home or in the clinic with or without mobility aids.
5. The subject is willing to accept treatment with a porcine based product and to undergo weekly compression wrapping.
6. The subject is medically stable, in the opinion of the investigator.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment

1. Index Ulcer Assessment:

   1. Penetrates down to muscle, tendon, or bone.
   2. Presence of another venous leg ulcer within 2 cm of the index ulcer
   3. Index ulcer determined to be due to a condition other than venous insufficiency.
   4. Exhibits overt clinical signs and symptoms of infection with cellulitis surrounding the wound margin.
   5. Known or suspected local skin malignancy to the index diabetic ulcer.
   6. Wound duration > one year without intermittent closure.
2. Prior therapies - Subjects receiving treatment with any of the following will not be eligible for enrollment:

   1. In the last 7 days - Negative pressure wound therapy (wound vac or SNaP®) of the index ulcer
   2. In the last 7 days - Hyperbaric oxygen (HBO) therapy
   3. In the last 30 days - Treatment with cytotoxic chemotherapy, application of topical steroids to the ulcer surface, or use of ≥ 14 days of immune-suppressants (including systemic corticosteroids); or subject is anticipated to require such medications during the course of the study
   4. In the last 30 days - study ulcer treatment with any advanced therapy, including, biomedical or topical growth factors, tissue engineered materials (e.g. Apligraf or Dermagraft), sterilized placental allografts (EpiFix, NovaFix, etc.), or other scaffold materials (e.g. OASIS® Wound Matrix, MatriStem Wound Matrix )
   5. In the last 8 weeks - Amputation or revascularization (surgical or stenting) to the affected leg
3. Subject criteria that will make subject ineligible for enrollment:

   1. Known hypersensitivity to porcine based products.
   2. Known osteomyelitis or active cellulitis requiring antimicrobial therapy at wound site.
   3. End stage renal disease requiring dialysis.
   4. Immune system disorders including Systemic Lupus Erythematosus (SLE), Acquired Immunodeficiency Syndrome (AIDS) or HIV
   5. Presence of any condition (including current drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol in the judgment of the Investigator.
   6. Pregnancy at enrollment or women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
   7. Subjects currently enrolled in this study. Concurrent enrollment in the study is prohibited.
   8. Subjects currently receiving radiation therapy or chemotherapy.
   9. Any pathology that would limit the blood supply and compromise healing or non-revascularizable surgical sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will consist of SerenaGroup® advanced wound care centers or affiliates that will enroll a minimum of 30 subjects.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound Area | 12 Weeks
  Assessment of ulcer area (percent area reduction from baseline)

SECONDARY OUTCOMES:
Time to complete wound closure | 12 Weeks
  Time to complete wound closure as defined by FDA.
Rate of wound closure | 12 Weeks
  Rate of wound closure as assessed by wound area measurements determined by weekly percent area reduction.
Adverse Events | 12 Weeks
  Incidence of adverse events
Reduction in pain | 12 Weeks
  Assessment of the pain level linked to the wound, using the validated PEG pain scale (0-10), with a higher score indicating more severe pain and pain-related interference with life and activities.

OTHER OUTCOMES:
Patient compliance with recommendations | 12 Weeks
  Patient compliance with behavioral treatment recommendations for the healing of venous leg ulceration. Treatment recomendations defined as multilayer compression therapy (as supplied by SerenaGroup®), with weekly assessments of effectiveness of multilayer compression with patient compliance.
App Usability | End of Study
  Assess ease of device using SUS questionnaire for WoundAlert smartphone application. To be completed by subject and provider
  The SUS scoring rule is as follows: (1) based on the level, each problem has a base score that ranges from 1-5, which corresponds to the range from "strongly disagree" to "strongly agree"; (2) the scores for questions 1, 3, 5, 7, and 9 are equal to the base score minus 1; the scores for questions 2, 4, 6, 8, and 10 are equal to five minus the base score; (3) the scores of the ten questions are added to obtain the total score of the questionnaire; and the questionnaire SUS score is the total score times 2.5. The SUS is represented as a percentage.
Bacterial Burden | 12 Weeks
  Reduction in bacterial burden as assessed by fluorescence imaging and polymerase chain reaction (PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- The Serena Group, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided